CLINICAL TRIAL: NCT05807529
Title: A Phase I-II, Dose-escalation, Double-blinded, Placebo-controlled, and Dose-finding Study to Evaluate the Safety and Efficacy of 2ccPA in Patients With Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Safety and Efficacy of 2ccPA in Patients With Symptomatic Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OEP-2PM102-201
Record Dates: First submitted 2022-12-29; First posted 2023-04-11 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — 2-carba-cyclic phosphatidic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2ccPA (Experimental): IP name: 2-carba-cyclic phosphatidic acid (2ccPA)
  Interventions: Drug: 2ccPA
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2ccPA — 2-carba-cyclic phosphatidic acid (2ccPA) is a first-in-class phospholipase autotaxin (ATX) inhibitor that may act as a disease-modifying drug and may relieve OA associated symptoms.
  Phase I: 2 dose cohorts (4800μg, 7200μg) single dose at Day 1
  Phase II: 3 dose cohorts (2400μg, 4800μg, 7200μg) multiple dose at Day 1, 15, 29
  Other Names: 2-carba-cyclic phosphatidic acid
  Arms: 2ccPA
Drug: Placebo — Phase I: 2 dose cohorts (4800μg, 7200μg) single dose at Day 1
  Phase II: 3 dose cohorts (2400μg, 4800μg, 7200μg) multiple dose at Day 1, 15, 29
  Arms: placebo

SUMMARY:
This phase I/II study aims to evaluate the safety of single doses of 2ccPA 4,800 μg and 7,200 μg (Phase I), as well as the safety and efficacy of multiple doses of 2ccPA (Phase II) in patients with osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease frequently associated with symptoms such as inflammation, stiffness, muscle weakness, joint swollen and joint pain. 2-carba-cyclic phosphatidic acid (2ccPA) is the derivative of natural occurring phospholipid mediator, cyclic phosphatidic acid (cPA). Previous studies suggested that 2ccPA inhibits inflammation and may relieve the pain caused by osteoarthritis. This phase I/II study aims to evaluate the safety of single doses of 2ccPA 4,800 μg and7,200 μg (Phase I), as well as the safety and efficacy of multiple doses of 2ccPA (Phase II) in patients with osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent from any patient capable of giving consent.
2. Male or female patients, 40 to 80 years of age.
3. Documented clinical diagnosis of symptomatic OA affecting at least one knee of a minimum of 6 months prior to screening.
4. The study knee has OA of Grade 2 to 3 severity based on the Kellgren Lawrence grading scale.
5. A score > 6 and < 16 out of 20 on the WOMAC pain subscale for the study knee.
6. Pain in the study knee for most of the 30 days (i.e., more than half of the days) prior to randomization.
7. Women of childbearing potential must agree to practice a medically acceptable contraceptive regimen from screening visit until at least 1 month after the study treatment and must have a negative pregnancy test no earlier than 72 hours prior to study treatment. Male subjects must agree to practice a medically acceptable contraceptive regimen (i.e., sterilization surgery, barrier method, abstention) from screening visit until at least 1 month after the study treatment.

Exclusion Criteria:

1. Patients with known or suspected hypersensitivity to 2ccPA or any of its excipients.
2. Use of intra-articular corticosteroids, hyaluronic acid, or other IA injection in the study knee within 3 months prior to study entry (randomization).
3. Use of chondroitin and/or glucosamine within 4 weeks prior to study entry (randomization).
4. Administered or requiring systemic or topical treatment of the study knee joint including immunosuppressive agents, anti-inflammatory drugs, steroids, or opioids for knee OA within 1 week prior to randomization. Acetaminophen (oral daily dose ≤ 3000 mg or topical use at any dose) can be taken up to 24 hours prior to randomization. For long-acting steroids (i.e., dexamethasone, betamethasone), subjects who received systemic treatment within 2 weeks before randomization will be excluded.
5. History of post-traumatic knee arthritis, or evidence of intra-articular bleeding of the study knee.
6. History of reiter's syndrome, gouty arthritis, systemic lupus erythematosus (SLE), sicca syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, lymphoma, arthritis associated with inflammatory bowel disease, sarcoidosis, amyloidosis or any other immune disease that based on investigators' discretion.
7. Periarticular inflammation from any cause, including referred pain, bursitis, tendonitis, soft tissue tenderness or acute pain from injury.
8. Subjects with clinical signs and symptoms of active knee infection or being treated for knee infection at screening.
9. Arthroscopic or open surgery on the study knee within 6 months prior to study entry (randomization).
10. Prior knee replacement on the study knee or planned knee replacement during the study period.
11. Subjects with meniscus tears that require repairment surgery or known anterior cruciate ligament rupture.
12. Subjects with known severe synovitis, synovium necrosis in the study knee joint.
13. Subjects with known malignancy.
14. Use of any chemotherapeutic or systemic immunosuppressant agents for inflammatory diseases within 6 months prior to study entry (randomization).
15. Current use of anticoagulants, including warfarin, heparin, low molecular weight heparin, dabigatran, or factor Xa inhibitors (rivaroxaban, apixaban, edoxaban, and betrixaban). Subject requiring routine use of low-dose aspirin for preventing thrombosis (≤ 100 mg/day) will not be excluded.
16. Abnormalities of laboratory parameters as described below will qualify for exclusion:

    * hemoglobin < 8 g/dL
    * total white blood cell count < lower limit of normal (LLN)
    * serum bilirubin/ alanine aminotransferase (ALT)/ aspartate aminotransferase AST > 2.5 times upper limit of normal (ULN)
    * serum creatinine > 2 times ULN
17. Pregnancy or lactation.
18. History of drug or alcohol dependence in the past 3 years.
19. Having known infection with HIV-1, active hepatitis B, or active hepatitis C. Patients who are inactive carriers of HBV or HCV can be enrolled if the subjects have stable baseline condition during the screening period.
20. Use of any investigational drug or participation in any drug study within 4 weeks prior to study entry (randomization).
21. Subjects unwilling or unable to comply with study procedures.
22. Any clinical condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk to participate in the study or confounds the ability to interpret data from the study as judged by the investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To define maximum tolerated dose (MTD) following the intra-articular (IA) administration of a single ascending dose (SAD) 2ccPA in patients with osteoarthritis of the knee. | 85 Days
To evaluate the safety of 2ccPA including incidence of adverse events (AEs) and serious adverse events (SAEs). | 85 Days
To evaluate the efficacy of multiple doses of 2ccPA vs placebo in terms of changes in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) on Day 85 | 85 Days
  The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with Osteoarthritis (OA) of the knee and hip, including pain (5 questions), stiffness (2 questions) and physical functioning (17 questions) of the joints. Each question is scored on a scale of 0-4, which corresponds to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).

SECONDARY OUTCOMES:
To evaluate the efficacy of 2ccPA vs placebo in terms of changes in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) on Day 15, 29, 57 and 168 | 85 Days
  WOMAC questionnaire consists of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), Physical Function (17 items). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
To evaluate the efficacy of 2ccPA vs placebo in terms of proportion of subjects with a 20% (WOMAC20), 50% (WOMAC50), and 70% (WOMAC70) improvement in the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) on Days 15, 29, 57, 85 and 168 | 168 Days
To evaluate the efficacy of 2ccPA vs placebo in terms of pain assessed by Numeric Rating Scale (NRS) on Days 15, 29, 57, 85 and 168. | 168 Days
  NRS is an 11-point numeric scale ranges from '0' indicating "no pain" to '10' indicating "extreme pain".
To evaluate the efficacy of 2ccPA vs placebo in terms of changes in Joint Space Narrowing (JSN) measured by x-ray on Day 168 | 168 Days
Maximum plasma concentration (Cmax) of 2ccPA | 168 Days
  Pharmacokinetic profile of 2ccPA
Time to maximum plasma concentration (Tmax) of 2ccPA | 168 Days
  Pharmacokinetic profile of 2ccPA
Area under plasma concentration-time curve (AUC0-infinity and AUC0-t) of 2ccPA | 168 Days
  Pharmacokinetic profile of 2ccPA
Apparent total body clearance (CL/F) of 2ccPA | 168 Days
  Pharmacokinetic profile of 2ccPA
Apparent volume of distribution (Vz/F) of 2ccPA | 168 Days
  Pharmacokinetic profile of 2ccPA
Elimination half-life (t1/2) of 2ccPA | 168 Days
  Pharmacokinetic profile of 2ccPA

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Cheng Chen, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan